CLINICAL TRIAL: NCT03338790
Title: A Phase 2 Study of Nivolumab in Combination With Either Rucaparib, Docetaxel, or Enzalutamide in Men With Castration-resistant Metastatic Prostate Cancer
Brief Title: An Investigational Immunotherapy Study of Nivolumab in Combination With Rucaparib, Docetaxel, or Enzalutamide in Metastatic Castration-resistant Prostate Cancer
Acronym: CheckMate 9KD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Clovis Oncology, Inc. (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9KD
Record Dates: First submitted 2017-11-08; First posted 2017-11-09 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; Docetaxel; enzalutamide; rucaparib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- nivolumab + rucaparib (Experimental): Specified dose on specified days
  Interventions: Biological: nivolumab; Drug: rucaparib
- nivolumab + docetaxel + prednisone (Experimental): Specified dose on specified days
  Interventions: Biological: nivolumab; Drug: docetaxel; Drug: prednisone
- nivolumab + enzalutamide (Experimental): Specified dose on specified days
  Interventions: Biological: nivolumab; Drug: enzalutamide

INTERVENTIONS:
Biological: nivolumab — Specified dose on specified days
  Other Names: BMS-936558, Opdivo
Drug: docetaxel — Specified dose on specified days
  Arms: nivolumab + docetaxel + prednisone
Drug: enzalutamide — Specified dose on specified days
  Arms: nivolumab + enzalutamide
Drug: rucaparib — Specified dose on specified days
  Arms: nivolumab + rucaparib
Drug: prednisone — Specified dose on specified days
  Arms: nivolumab + docetaxel + prednisone

SUMMARY:
The purpose of this study is to assess safety and efficacy of nivolumab in combination with rucaparib, docetaxel, or enzalutamide in participants with castration-resistant prostate cancer that has spread.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate
* Evidence of stage IV disease on previous bone, CT, and/or MRI scan
* Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy
* Mandatory plasma and fresh or archival tumor tissue must be submitted

Exclusion Criteria:

* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast
* Participants with active brain metastases
* Participants must have recovered from the effects of major surgery requiring general anesthesia or significant traumatic injury at least 14 days before treatment arm assignment

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 292 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (19):
  - Local Institution - 0036, Daphne, Alabama
  - Local Institution - 0010, Rancho Mirage, California
  - Local Institution - 0049, New Haven, Connecticut
  - Local Institution - 0037, Miami, Florida
  - Local Institution - 0009, Marietta, Georgia
  - Local Institution - 0065, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Local Institution - 0040, Rockville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Local Institution - 0012, Detroit, Michigan
  - Local Institution - 0069, Jackson, Mississippi
  - Local Institution - 0011, St Louis, Missouri
  - Local Institution - 0035, Omaha, Nebraska
  - Local Institution - 0038, Albany, New York
  - Local Institution - 0068, New York, New York
  - Local Institution - 0041, Durham, North Carolina
  - Local Institution - 0024, Portland, Oregon
  - Local Institution - 0053, Allentown, Pennsylvania
  - Local Institution - 0039, Fairfax, Virginia
- Argentina (5):
  - Local Institution - 0052, CABA, Buenos Aires
  - Local Institution - 0042, Capital Federal, Buenos Aires
  - Local Institution - 0062, Villa Siburu, Córdoba Province
  - Local Institution - 0044, Buenos Aires, Distrito Federal
  - Local Institution - 0043, CABA
- Australia (6):
  - Local Institution - 0015, Camperdown, New South Wales
  - Local Institution - 0017, Westmead, New South Wales
  - Local Institution - 0014, South Brisbane, Queensland
  - Local Institution - 0016, Elizabeth Vale, South Australia
  - Local Institution - 0050, Clayton, Victoria
  - Local Institution - 0013, Heidelberg, Victoria
- Brazil (9):
  - Local Institution - 0020, Belo Horizonte, Minas Gerais
  - Local Institution - 0074, Belo Horizonte, Minas Gerais
  - Local Institution - 0075, Curitiba, Paraná
  - Local Institution - 0019, Rio de Janeiro, Rio de Janeiro
  - Local Institution - 0018, Ijuí, Rio Grande do Sul
  - Local Institution - 0021, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0022, Campinas, São Paulo
  - Local Institution - 0073, São Paulo, São Paulo
  - Local Institution - 0071, São Paulo, São Paulo
- Canada (5):
  - Local Institution - 0067, Kelowna, British Columbia
  - Local Institution - 0059, Moncton, New Brunswick
  - Local Institution - 0055, Hamilton, Ontario
  - Local Institution - 0066, Montreal, Quebec
  - Local Institution - 0056, Québec, Quebec
- Chile (2):
  - Local Institution - 0051, Viña del Mar, Región de Valparaíso
  - Local Institution - 0034, Santiago, Santiago Metropolitan
- Colombia (2):
  - Local Institution - 0027, Montería, Departamento de Córdoba
  - Local Institution - 0026, Medellín
- France (5):
  - Local Institution - 0033, Besançon
  - Local Institution - 0032, Clermont-Ferrand
  - Local Institution - 0031, Lyon
  - Local Institution - 0030, Marseille
  - Local Institution - 0029, Villejuif
- Germany (6):
  - Local Institution - 0001, Essen
  - Local Institution - 0006, Göttingen
  - Local Institution - 0004, Heidelberg
  - Local Institution - 0002, Jena
  - Local Institution - 0007, Koblenz
  - Local Institution - 0064, München
- Mexico (4):
  - Local Institution - 0054, León, Guanajuato
  - Local Institution - 0061, Guadalajara, Jalisco
  - Local Institution - 0048, Guadalajara, Jalisco
  - Local Institution - 0025, Culiacán, Sinaloa
- Spain (3):
  - Local Institution - 0045, Madrid
  - Local Institution - 0046, Pamplona
  - Local Institution - 0047, Seville

REFERENCES:
- [Derived] Fizazi K, Retz M, Petrylak DP, Goh JC, Perez-Gracia J, Lacombe L, Zschabitz S, Burotto M, Mahammedi H, Gravis G, Bastos DA, McCune SL, Vazquez Limon JC, Kwan EM, Castellano D, Flechon A, Saad F, Grimm MO, Shaffer DR, Armstrong AJ, Bhagavatheeswaran P, Amin NP, Unsal-Kacmaz K, Wang X, Li J, Loehr A, Pachynski RK. Nivolumab plus rucaparib for metastatic castration-resistant prostate cancer: results from the phase 2 CheckMate 9KD trial. J Immunother Cancer. 2022 Aug;10(8):e004761. doi: 10.1136/jitc-2022-004761. PMID 35977756
- [Derived] Fizazi K, Gonzalez Mella P, Castellano D, Minatta JN, Rezazadeh Kalebasty A, Shaffer D, Vazquez Limon JC, Sanchez Lopez HM, Armstrong AJ, Horvath L, Bastos DA, Amin NP, Li J, Unsal-Kacmaz K, Retz M, Saad F, Petrylak DP, Pachynski RK. Nivolumab plus docetaxel in patients with chemotherapy-naive metastatic castration-resistant prostate cancer: results from the phase II CheckMate 9KD trial. Eur J Cancer. 2022 Jan;160:61-71. doi: 10.1016/j.ejca.2021.09.043. Epub 2021 Nov 18. PMID 34802864
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 292 participants treated
Groups:
- Arm A1: Nivolumab 480 mg IV Q4W + Rucaparib 600 mg PO BID for participants who have at lease 1 but no more than 2 prior chemotherapy regimens
- Arm A2: Nivolumab 480 mg IV Q4W + Rucaparib 600 mg PO BID for participants who have not received prior chemotherapy regimen
- Arm B: Nivolumab 360 mg IV Q3W + Docetaxel 75 mg/m2 IV Q3W + Prednisone 5 mg PO BID
- Arm C: Nivolumab 480 mg IV Q4W + Enzalutamide 160 mg PO QD
Period: Overall Study
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Started (Started = Treated) | 88 | 71 | 84 | 49
Completed | 0 | 3 | 1 | 0
Not Completed | 88 | 68 | 83 | 49
Not completed — Disease Progression | 65 | 46 | 54 | 42
Not completed — Study Drug Toxicity | 12 | 8 | 14 | 0
Not completed — Death | 2 | 1 | 1 | 0
Not completed — Adverse Event unrelated to Study Drug | 4 | 4 | 6 | 4
Not completed — Participant request to discontinue study treatment | 4 | 3 | 3 | 1
Not completed — Poor/non-compliance | 0 | 1 | 0 | 0
Not completed — Participant withdrew consent | 1 | 0 | 1 | 1
Not completed — Other reasons | 0 | 5 | 1 | 1
Not completed — Maximum clinical benefit | 0 | 0 | 1 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C | Total
Number analyzed (Participants) | 88 | 71 | 84 | 49 | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (8.3) | 70.7 (9.7) | 70.3 (7.6) | 69.8 (8.0) | 69.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 88 | 71 | 84 | 49 | 292
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 8 | 2 | 15
  White | 72 | 64 | 70 | 42 | 248
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 5 | 5 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Per Prostate Cancer Clinical Trials Working Group 3 (ORR-PCWG3)
Description: Objective response rate per prostate cancer clinical trials working group 3 (ORR-PCWG3) for target lesions and assessed by MRI is the percentage of participants who have a confirmed complete or partial best overall response (BOR) per PCWG3 among treated participants who have measurable disease
Time Frame: Up to approximately 36 months
Population: All response evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 58 | 39 | 45 | 18
Percentage of participants
  Overall | 10.3 [3.9 to 21.2] | 15.4 [5.9 to 30.5] | 40.0 [25.7 to 55.7] | 11.1 [1.4 to 34.7]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 29 | 20 | 19 | 5
  Homologous Recombination Deficiency (HRD+) | 17.2 [5.8 to 35.8] | 25.0 [8.7 to 49.1] | 36.8 [16.3 to 61.6] | 20.0 [0.5 to 71.6]

2. Primary Outcome: Prostate-Specific Antigen Response Rate (RR-PSA)
Description: Prostate-specific antigen response rate (RR-PSA) is the percentage of treated participants with a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result
Time Frame: Up to approximately 36 months
Population: All treated participants with baseline and at least one post-baseline PSA assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 84 | 66 | 81 | 44
Percentage of participants
  Overall | 11.9 [5.9 to 20.8] | 27.3 [17.0 to 39.6] | 46.9 [35.7 to 58.3] | 34.1 [20.5 to 49.9]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 44 | 31 | 34 | 10
  Homologous Recombination Deficiency (HRD+) | 18.2 [8.2 to 32.7] | 41.9 [24.5 to 60.9] | 50.0 [32.4 to 67.6] | 50.0 [18.7 to 81.3]

3. Secondary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: Radiographic progress-free survival (rPFS) is the time between treatment initiation and the first date of documented progression or death due to any cause, whichever occurs first assessed by the investigator per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)
Time Frame: Up to approximately 84 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 71 | 84 | 49
Months
  Overall | 4.60 [3.68 to 5.72] | 8.15 [5.59 to 10.97] | 9.20 [8.25 to 11.47] | 5.75 [3.81 to 9.33]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 45 | 34 | 35 | 12
  Homologous Recombination Deficiency (HRD+) | 5.59 [3.68 to 8.08] | 11.01 [6.74 to 12.02] | 10.45 [8.44 to 12.88] | 8.48 [3.78 to NA] — Upper limit not reached due to too few events

4. Secondary Outcome: Time to Response Per Prostate Cancer Clinical Trials Working Group 3 (TTR-PCWG3)
Description: Time to response per prostate cancer clinical trials working group 3 (TTR-PCWG3) is the time from treatment initiation to the date of the first documented complete response (CR) or partial response (PR) per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)
Time Frame: Up to approximately 84 months
Population: All response evaluable participants (CR or PR)
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 7 | 6 | 21 | 2
Months
  Overall | 1.94 [1.6 to 5.1] | 1.95 [1.8 to 11.0] | 1.94 [1.6 to 8.3] | 1.9 [1.9 to 1.9]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 6 | 5 | 9 | 1
  Homologous Recombination Deficiency (HRD+) | 2.76 [1.6 to 5.1] | 2.07 [1.8 to 11.0] | 2.04 [1.8 to 8.3] | 1.9 [1.9 to 1.9]

5. Secondary Outcome: Duration of Response Per Prostate Cancer Clinical Trials Working Group 3 (DOR-PCWG3)
Description: Duration of response per prostate cancer clinical trials working group 3 (DOR-PCWG3) is the time between the date of first response (complete response/partial response per PCWG3) to the date of first documented radiographic progression per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) or death due to any cause
Time Frame: Up to approximately 84 months
Population: All response evaluable participants (CR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 7 | 6 | 21 | 2
Months
  Overall | NA [3.45 to NA] — Median and upper limit not reached due to too few events | 7.10 [3.78 to NA] — Upper limit not reached due to too few events | 7.21 [6.47 to 12.35] | NA [9.23 to NA] — Median and upper limit not reached due to too few events
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 6 | 5 | 9 | 1
  Homologous Recombination Deficiency (HRD+) | NA [3.45 to NA] — Median and upper limit not reached due to too few events | 7.10 [3.78 to NA] — Upper limit not reached due to too few events | 7.43 [6.44 to 13.86] | NA [NA to NA] — Median and upper limit not reached due to too few events

6. Secondary Outcome: Prostate-Specific Antigen Time to Progression (TTP-PSA)
Description: Prostate-specific antigen time to progression (TTP-PSA) is the time between treatment initiation to the date of PSA progression per prostate cancer clinical trials working group 3 (PCWG3)
Time Frame: Up to approximately 84 months
Population: All PSA response evaluable participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 85 | 66 | 81 | 44
Months
  Overall | 3.78 [2.83 to 6.47] | 3.45 [2.83 to 6.21] | 8.67 [7.16 to 10.35] | 3.09 [2.79 to 6.37]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 44 | 32 | 34 | 10
  Homologous Recombination Deficiency (HRD+) | 6.47 [3.78 to 9.63] | 10.25 [4.63 to 13.77] | 8.64 [7.16 to 10.58] | 5.55 [2.73 to 8.28]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is the time between treatment initiation and the date of death from any cause. For participants who are alive, their survival time will be censored at the last date that they were known to be alive. OS will be censored for participants at the date of treatment initiation if they had no follow-up
Time Frame: Up to approximately 84 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 71 | 84 | 49
Months
  Overall | 13.96 [10.35 to 15.77] | 20.24 [13.54 to 22.90] | 18.17 [15.15 to 25.49] | 17.41 [12.98 to 24.15]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 45 | 34 | 35 | 12
  Homologous Recombination Deficiency (HRD+) | 15.15 [11.40 to 18.20] | 23.00 [13.54 to 29.27] | 19.35 [13.54 to 27.20] | 24.97 [9.10 to 45.50]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of Participants with any grade adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and immune-mediated AEs using the Common Toxicity Criteria Grade for Adverse Events (CTCAE V4)
Time Frame: From first dose to up to 30 days post last dose (Up to 82 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 71 | 84 | 49
Participants
  Adverse Events (AEs) | 88 | 71 | 83 | 49
  Serious Adverse Events (SAEs) | 49 | 37 | 41 | 20
  AEs leading to discontinuation | 47 | 31 | 37 | 17
  Immune-mediated AEs (Pneumonitis) | 1 | 2 | 9 | 0
  Immune-mediated AEs (Diarrhea/Colitis) | 3 | 4 | 2 | 0
  Immune-mediated AEs (Hepatitis) | 8 | 6 | 1 | 2
  Immune-mediated AEs (Nephritis/Renal Dysfunction) | 0 | 3 | 0 | 0
  Immune-mediated AEs (Rash) | 6 | 5 | 7 | 10
  Immune-mediated AEs (Hypersensitivity) | 0 | 0 | 0 | 3
  Immune-mediated AEs (Adrenal insufficiency) | 1 | 0 | 0 | 0
  Immune-mediated AEs (Hypothyroidism/Thyroiditis) | 7 | 6 | 3 | 5
  Immune-mediated AEs (Hyperthyroidism) | 2 | 1 | 2 | 0
  Immune-mediated AEs (Hypophysitis) | 0 | 0 | 1 | 0
  Immune-mediated AEs (Diabetes Mellitus) | 0 | 1 | 0 | 1

9. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause.
Time Frame: Up to 84 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 71 | 84 | 49
Participants | 79 | 66 | 76 | 47

10. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants with laboratory abnormalities in specific liver tests based on SI conventional units to assess the overall safety and tolerability of BMS-986213 in combination with chemotherapy vs. Nivolumab in combination with chemotherapy. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * ALP > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
Time Frame: From first dose to up to 30 days post last dose (up to 82 months)
Population: All treated participant with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Number; unit: Participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 69 | 84 | 48
Participants
  ALT or AST > 3xULN | 19 | 23 | 6 | 4
  ALT or AST > 5xULN | 11 | 15 | 3 | 3
  ALT or AST > 10xULN | 2 | 5 | 1 | 0
  ALT or AST > 20xULN | 0 | 1 | 1 | 0
  TOTAL BILIRUBIN > 2xULN | 3 | 1 | 1 | 0
  ALP > 1.5xULN | 49 | 34 | 35 | 22
  Concurrent ALT or AST elevation > 3xULN with total Bilirubin > 1.5xULN within one day | 3 | 1 | 0 | 1
  Concurrent ALT or AST elevation > 3xULN with total Bilirubin > 1.5xULN within 30 days | 4 | 1 | 0 | 1
  Concurrent ALT or AST elevation > 3xULN with total Bilirubin > 2xULN within one day | 2 | 1 | 0 | 0
  Concurrent ALT or AST elevation > 3xULN with total Bilirubin > 2xULN within 30 days | 2 | 1 | 0 | 0

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of participants with laboratory abnormalities in specific thyroid tests based on US conventional units. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * TSH value > ULN and
  * with baseline TSH value <= ULN
  * with at least one FT3/FT4 test value < LLN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values >= LLN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test.
  * TSH < LLN and
  * with baseline TSH value >= LLN
  * with at least one FT3/FT4 test value > ULN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values <= ULN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test
Time Frame: From first dose to up to 30 days post last dose (Up to 82 months)
Population: All treated participants with thyroid stimulating hormone (TSH) abnormality
Measure: Number; unit: Participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 71 | 84 | 49
Participants
  TSH > ULN | 23 | 17 | 12 | 17
  TSH > ULN with TSH <= ULN at baseline | 18 | 12 | 7 | 12
  TSH > ULN with at least one FT3/FT4 test value < LLN | 10 | 6 | 7 | 5
  TSH > ULN with all other FT3/FT4 test values >= LLN | 11 | 9 | 3 | 9
  TSH > ULN with FT3/FT4 test missing | 2 | 2 | 2 | 3
  TSH < LLN | 17 | 12 | 25 | 8
  TSH < LLN with TSH >= LLN at baseline | 14 | 11 | 19 | 8
  TSH < LLN with at least one FT3/FT4 test value > ULN | 6 | 5 | 2 | 7
  TSH < LLN with all other FT3/FT4 test values <= ULN | 8 | 4 | 11 | 0
  TSH < LLN with FT3/FT4 test missing | 3 | 3 | 12 | 1

12. Secondary Outcome: Number of Participants With Laboratory Values Change From Baseline
Description: Number of participants changed from baseline in laboratory values of worst toxicity grade (grade 0= wnl, grade 1= mild, grade 2= moderate, grade 3= severe) based on US conventional units by cohort
Time Frame: From first dose to up to 30 days post last dose (Up to 82 months)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 88 | 71 | 84 | 49
Participants
  Hemoglobin Grade 0: number analyzed (Participants) | 24 | 23 | 31 | 12
  Hemoglobin Grade 0 | 23 | 21 | 30 | 8
  Hemoglobin Grade 1: number analyzed (Participants) | 55 | 41 | 48 | 30
  Hemoglobin Grade 1 | 38 | 28 | 23 | 13
  Hemoglobin Grade 2: number analyzed (Participants) | 9 | 5 | 4 | 4
  Hemoglobin Grade 2 | 8 | 3 | 2 | 2
  Platelet Grade 0: number analyzed (Participants) | 82 | 66 | 79 | 43
  Platelet Grade 0 | 34 | 32 | 10 | 13
  Platelet Grade 1: number analyzed (Participants) | 6 | 2 | 4 | 3
  Platelet Grade 1 | 4 | 1 | 0 | 0
  Leukocytes Grade 0: number analyzed (Participants) | 76 | 61 | 76 | 41
  Leukocytes Grade 0 | 39 | 35 | 30 | 13
  Leukocytes Grade 1: number analyzed (Participants) | 11 | 7 | 6 | 5
  Leukocytes Grade 1 | 10 | 6 | 3 | 3
  Leukocytes Grade 2: number analyzed (Participants) | 1 | 1 | 1 | 0
  Leukocytes Grade 2 | 1 | 0 | 1 |
  Lymphocytes Grade 0: number analyzed (Participants) | 44 | 48 | 55 | 24
  Lymphocytes Grade 0 | 24 | 30 | 28 | 14
  Lymphocytes Grade 1: number analyzed (Participants) | 13 | 10 | 4 | 4
  Lymphocytes Grade 1 | 11 | 8 | 1 | 2
  Lymphocytes Grade 2: number analyzed (Participants) | 8 | 4 | 12 | 8
  Lymphocytes Grade 2 | 3 | 3 | 6 | 3
  Lymphocytes Grade 3: number analyzed (Participants) | 4 | 2 | 6 | 0
  Lymphocytes Grade 3 | 1 | 0 | 0 |
  Neutrophil Grade 0: number analyzed (Participants) | 82 | 63 | 81 | 45
  Neutrophil Grade 0 | 35 | 26 | 38 | 7
  Neutrophil Grade 1: number analyzed (Participants) | 4 | 6 | 1 | 0
  Neutrophil Grade 1 | 3 | 4 | 1 |
  Neutrophil Grade 2: number analyzed (Participants) | 2 | 0 | 0 | 1
  Neutrophil Grade 2 | 1 |  |  | 1
  Alkaline Phosphatase Grade 0: number analyzed (Participants) | 47 | 51 | 41 | 27
  Alkaline Phosphatase Grade 0 | 25 | 34 | 13 | 8
  Alkaline Phosphatase Grade 1: number analyzed (Participants) | 28 | 10 | 30 | 14
  Alkaline Phosphatase Grade 1 | 14 | 4 | 13 | 6
  Alkaline Phosphatase Grade 2: number analyzed (Participants) | 12 | 3 | 9 | 2
  Alkaline Phosphatase Grade 2 | 9 | 1 | 3 | 0
  Alkaline Phosphatase Grade 3: number analyzed (Participants) | 1 | 5 | 3 | 3
  Alkaline Phosphatase Grade 3 | 1 | 3 | 0 | 0
  Aspartate Aminotransferase Grade 0: number analyzed (Participants) | 71 | 64 | 74 | 37
  Aspartate Aminotransferase Grade 0 | 52 | 49 | 16 | 9
  Aspartate Aminotransferase Grade 1: number analyzed (Participants) | 17 | 5 | 8 | 9
  Aspartate Aminotransferase Grade 1 | 5 | 4 | 6 | 4
  Alanine Aminotransferase Grade 0: number analyzed (Participants) | 82 | 63 | 78 | 42
  Alanine Aminotransferase Grade 0 | 48 | 48 | 13 | 4
  Alanine Aminotransferase Grade 1: number analyzed (Participants) | 6 | 6 | 5 | 4
  Alanine Aminotransferase Grade 1 | 4 | 3 | 3 | 1
  Bilirubin Grade 0: number analyzed (Participants) | 87 | 69 | 83 | 45
  Bilirubin Grade 0 | 16 | 12 | 2 | 3
  Bilirubin Grade 1: number analyzed (Participants) | 1 | 0 | 0 | 1
  Bilirubin Grade 1 | 1 |  |  | 0
  Creatinine Grade 0: number analyzed (Participants) | 77 | 62 | 74 | 43
  Creatinine Grade 0 | 31 | 30 | 13 | 3
  Creatinine Grade 1: number analyzed (Participants) | 11 | 7 | 9 | 3
  Creatinine Grade 1 | 7 | 5 | 5 | 2

13. Post Hoc Outcome: Objective Response Rate Per Prostate Cancer Clinical Trials Working Group 3 (ORR-PCWG3) - Extended Collection
Description: as for outcome 1
Time Frame: Up to approximately 82 months
Population: All response evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 58 | 39 | 45 | 18
Percentage of participants
  Overall | 12.1 [5.0 to 23.3] | 15.4 [5.9 to 30.5] | 40.0 [25.7 to 55.7] | 11.1 [1.4 to 34.7]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 29 | 20 | 19 | 5
  Homologous Recombination Deficiency (HRD+) | 20.7 [8.0 to 39.7] | 25.0 [8.7 to 49.1] | 36.8 [16.3 to 61.6] | 20.0 [0.5 to 71.6]

14. Post Hoc Outcome: Prostate-Specific Antigen Response Rate (RR-PSA) - Extended Collection
Description: as for outcome 2
Time Frame: Up to approximately 82 months
Population: All response evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A1 | Arm A2 | Arm B | Arm C
Number analyzed (Participants) | 85 | 66 | 81 | 44
Percentage of participants
  Overall | 11.8 [5.8 to 20.6] | 28.8 [18.3 to 41.3] | 46.9 [35.7 to 58.3] | 34.1 [20.5 to 49.9]
  Homologous Recombination Deficiency (HRD+): number analyzed (Participants) | 44 | 32 | 34 | 10
  Homologous Recombination Deficiency (HRD+) | 18.2 [8.2 to 32.7] | 43.8 [26.4 to 62.3] | 50.0 [32.4 to 67.6] | 50.0 [18.7 to 81.3]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 84 months). SAEs and Other AEs were assessed from first dose to 100 days post the last dose (up to approximately 84 months).
Groups:
- Arm A1: Nivolumab 480 mg and Rucaparib 600 mg: Nivolumab 480 mg IV Q4W + Rucaparib 600 mg PO BID for participants who have at lease 1 but no more than 2 prior chemotherapy regimens
- Arm A2: Nivolumab 480 mg and Rucaparib 600 mg: Nivolumab 480 mg IV Q4W + Rucaparib 600 mg PO BID for participants who have not received prior chemotherapy regimen
- Arm B: Nivolumab 360 mg and Docetaxel 75 mg/m2: Nivolumab 360 mg IV Q3W + Docetaxel 75 mg/m2 IV Q3W + Prednisone 5 mg PO BID
- Arm C: Nivolumab 480 mg and Enzalutamide 160 mg: Nivolumab 480 mg IV Q4W + Enzalutamide 160 mg PO QD
Arm/Group | Arm A1: Nivolumab 480 mg and Rucaparib 600 mg | Arm A2: Nivolumab 480 mg and Rucaparib 600 mg | Arm B: Nivolumab 360 mg and Docetaxel 75 mg/m2 | Arm C: Nivolumab 480 mg and Enzalutamide 160 mg
All-Cause Mortality (participants affected / at risk) | 79/88 | 66/71 | 76/84 | 47/49
Serious Adverse Events (participants affected / at risk) | 53/88 | 45/71 | 50/84 | 25/49
Other Adverse Events (participants affected / at risk) | 87/88 | 70/71 | 83/84 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Nivolumab 480 mg and Rucaparib 600 mg (N=88) | Arm A2: Nivolumab 480 mg and Rucaparib 600 mg (N=71) | Arm B: Nivolumab 360 mg and Docetaxel 75 mg/m2 (N=84) | Arm C: Nivolumab 480 mg and Enzalutamide 160 mg (N=49)
Anaemia (Blood and lymphatic system disorders) | 8 | 4 | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 4 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Asthenia (General disorders and administration site conditions) | 0 | 0 | 2 | 1
Death (General disorders and administration site conditions) | 0 | 0 | 1 | 0
Fatigue (General disorders and administration site conditions) | 2 | 1 | 1 | 0
General physical health deterioration (General disorders and administration site conditions) | 3 | 1 | 0 | 0
Malaise (General disorders and administration site conditions) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders and administration site conditions) | 0 | 0 | 1 | 0
Pain (General disorders and administration site conditions) | 0 | 0 | 2 | 0
Pyrexia (General disorders and administration site conditions) | 2 | 1 | 1 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis orbital (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 9 | 6 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 4 | 3 | 1
Septic shock (Infections and infestations) | 1 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 1
Urosepsis (Infections and infestations) | 2 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular anastomosis aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 2 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 9 | 8 | 7
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Device occlusion (Product issues) | 1 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 2 | 1 | 1
Autoimmune nephritis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureteric compression (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinoma (Renal and urinary disorders) | 0 | 0 | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cutaneous sarcoidosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Lymphatic fistula (Vascular disorders) | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Nivolumab 480 mg and Rucaparib 600 mg (N=88) | Arm A2: Nivolumab 480 mg and Rucaparib 600 mg (N=71) | Arm B: Nivolumab 360 mg and Docetaxel 75 mg/m2 (N=84) | Arm C: Nivolumab 480 mg and Enzalutamide 160 mg (N=49)
Anaemia (Blood and lymphatic system disorders) | 32 | 30 | 25 | 15
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 14 | 4 | 14 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 8 | 2 | 3
Hypothyroidism (Endocrine disorders) | 7 | 5 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 9 | 5 | 11 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 4 | 1
Constipation (Gastrointestinal disorders) | 26 | 18 | 21 | 10
Diarrhoea (Gastrointestinal disorders) | 29 | 21 | 42 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 4 | 3
Nausea (Gastrointestinal disorders) | 46 | 35 | 36 | 17
Vomiting (Gastrointestinal disorders) | 30 | 18 | 14 | 5
Asthenia (General disorders and administration site conditions) | 24 | 12 | 17 | 11
Chills (General disorders and administration site conditions) | 4 | 6 | 9 | 1
Fatigue (General disorders and administration site conditions) | 36 | 26 | 41 | 21
Mucosal inflammation (General disorders and administration site conditions) | 8 | 1 | 6 | 1
Oedema peripheral (General disorders and administration site conditions) | 17 | 15 | 20 | 10
Pain (General disorders and administration site conditions) | 6 | 2 | 3 | 7
Pyrexia (General disorders and administration site conditions) | 15 | 7 | 13 | 4
Bronchitis (Infections and infestations) | 5 | 1 | 5 | 0
Pneumonia (Infections and infestations) | 6 | 6 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 5 | 0
Urinary tract infection (Infections and infestations) | 5 | 3 | 6 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 6 | 2
Alanine aminotransferase increased (Investigations) | 16 | 21 | 5 | 4
Aspartate aminotransferase increased (Investigations) | 15 | 21 | 4 | 7
Blood alkaline phosphatase increased (Investigations) | 8 | 9 | 4 | 5
Blood creatinine increased (Investigations) | 8 | 20 | 5 | 2
Neutrophil count decreased (Investigations) | 0 | 3 | 6 | 0
Platelet count decreased (Investigations) | 4 | 6 | 0 | 1
Transaminases increased (Investigations) | 3 | 4 | 2 | 1
Weight decreased (Investigations) | 9 | 7 | 6 | 5
Decreased appetite (Metabolism and nutrition disorders) | 29 | 21 | 25 | 14
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 6 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 4 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 11 | 20 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 11 | 25 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 7 | 8 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 5 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 6 | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 7 | 10 | 11
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4
Dizziness (Nervous system disorders) | 7 | 6 | 17 | 6
Dysgeusia (Nervous system disorders) | 11 | 9 | 12 | 6
Headache (Nervous system disorders) | 8 | 6 | 10 | 6
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 23 | 2
Paraesthesia (Nervous system disorders) | 2 | 3 | 3 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 5 | 0
Syncope (Nervous system disorders) | 0 | 1 | 3 | 3
Depression (Psychiatric disorders) | 2 | 6 | 2 | 4
Insomnia (Psychiatric disorders) | 8 | 6 | 9 | 8
Acute kidney injury (Renal and urinary disorders) | 5 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 7 | 3 | 5 | 1
Urinary retention (Renal and urinary disorders) | 3 | 3 | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 11 | 21 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 20 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 8 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 28 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 5 | 3 | 4
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4 | 1 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 11 | 6 | 9
Rash (Skin and subcutaneous tissue disorders) | 10 | 9 | 16 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 0
Hypertension (Vascular disorders) | 5 | 3 | 5 | 4
Hypotension (Vascular disorders) | 7 | 6 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03338790/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03338790/SAP_001.pdf